CLINICAL TRIAL: NCT04657653
Title: Hyperbaric Oxygen Therapy Versus Core Decompression Augmented With Bone Substitute in Pre Collapse of Avascular Necrosis of Femoral Head
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Isam Moghamis, medical resident, Hamad Medical Corporation
Other Study IDs: MRC/140/2017
Record Dates: First submitted 2020-11-25; First posted 2020-12-08 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: AVN
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: core decompression — :The procedure was performed under general anesthesia with the aid of image intensifier. All patients were positioned in supine position on a fracture table. The core decompression was performed using the direct lateral approach with 2 cm skin incision. A fluoroscope guided large single drill with 8 mm diameter over a guide wire was used to remove the necrotic tissues from the femur head through the lateral cortex distal to trochanteric tubercle. After the removal of the core necrotic bone, the track was filled with 5 ml synthetic bone paste substitute (tricalcium phosphate) and an intraoperative fluoroscope was used to confirm the adequacy of the decompression and grafting.
  Other Names: hyperbaric oxygen therapy

SUMMARY:
Introduction: osteonecrosis of the femoral head is a potentially crippling disorder, which mainly affects the young adults. Core decompression has been used for the treatment of the osteonecrosis of the femur head since was published by Ficat and albert, and by HUNGERFORD and Lennox. hyperbaric oxygen therapy is a suggestive joint preserving treatment for symptomatic prolapse stage of osteonecrosis of the femur head.

Aims and objectives: to compare the clinical (functional) outcome of core decompression versus hyperbaric oxygen therapy in pre collapse stages of idiopathic avascular necrosis of the femur head.

Material and methods: Mixed Retrospective and prospective study for all case of pre collapse of avascular necrosis of femoral head(AVNHF) underwent either hyperbaric oxygen therapy or Core decompression augmented with bone substitute in HAMAD General Hospital

Anticipated outcome: Hyperbaric oxygen treatment associated with better outcomes at preserving the joint and associated with less complications than surgery

DETAILED DESCRIPTION:
Methods Data were collected retrospectively from the medical records from 23 patients, between January 2010 and December 2018. The data for patient's demographic (age, gender, body metabolic index (BMI) comorbidities, risk factors for avascular necrosis (AVN), (diabetes mellitus (DM), hypertension (HTN), alcoholic, smoking, steroid used, sickle cell disease, chemo or radiation therapy), pre- and post- treatment radiological stage (Steinberg's classification) [15],functional outcome (oxford hip score and SF 12), complications and need for further surgical intervention or Total Hip Arthroplasty (THA) were collected.

Patients who were 18 years old or more, with non- traumatic AVN in pre-collapse stage (stage 1 or 2 Steinberg)[15] that was confirmed by MRI and underwent either hyperbaric oxygen therapy or core decompression with bone substitute augmentation with a minimum one year of follow up were included.

Patient with traumatic AVN, advanced stages of AVN (stages 3, 4 and 5), core decompression without bone graft, combined therapy, other hip procedures and less than one year follow up were excluded from the study.

Writing Informed consent was obtained from all patients and they were interviewed through their regular clinical follow up with a minimum of 1-year follow up after the treatment. The clinical outcome was measured using Oxford hip score(OHS) and short form 12 (SF12) for both groups, the forms were used in two languages Arabic and English, the Arabic form was translated through the institutional medical research center by a certified translator.

Radiological progression of AVN stage was assessed by comparing radiographs before and after treatment. All radiographs and MRI images were reviewed and certified musculoskeletal radiologist did staging.

Satisfactory clinical outcome was defined as OHS score of more than 30 and no further surgical interventions. Radiological progression was identified with more advanced stages in post treatment radiographs.

Core Decompression surgical procedure:

Data analysis Descriptive statistics were used to summarize the patients' demographic, comorbidities and radiological measurements. Chi-square test and Fisher Exact test were used to express the associations between two or more qualitative variables whereas unpaired Student t test was used to compare the quantitative data (Oxford Hip Score & SF12) between the two groups. Frequency (percentage) and mean ± standard deviation (SD) or median and range were used as appropriate for categorical and continuous values. The result was considered statistically significant if P value ≤.05. All statistical analyses were done using statistical packages SPSS 23.0 (SPSS Inc. Chicago, IL) and Epi information technology (InfoTM) 2000 (Centers for Disease Control and Prevention, Atlanta, GA)

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more,
* non- traumatic AVN stages 2 (Steinberg)
* pre treatment MRI
* underwent either hyperbaric oxygen therapy or core decompression with bone substitute augmentation
* minimum one year of follow up were included

Exclusion Criteria:

* traumatic AVN,
* other stages of AVN (stages 1, 3, 4 and 5),
* core decompression without bone graft,
* combined therapy, other hip procedures
* less than one year follow up were excluded from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 19 patients with 23 pre-collapsed stage 2 non-traumatic AVN of femoral head were included, 12 (52.2%) in core CD and 11 (47.8%) in HBO group with average of 39.5±13 sessions.
  9 (47.3%) males, 10 (52.7%) females, the average age was 35.2±9.8 years with average BMI 27.3±4.3 and follow up was 34.2±18.4 months.
  Risk factors was observed in 6 cases on steroid, 4 smokers, 1 DM, 3 sickle cell disease, 2 alcoholics, and 7 cases with no risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
compare the functional and radiological outcomes of the hyperbaric oxygen therapy (HBO) versus core decompression (CD) in pre-collapsed stage II of non-traumatic AVN of the femoral head. | between January 2010 and December 2018
  comparing the oxford hip score and short form 12 score between patient who underwent core decompression and patients who underwent hyperbaric oxygen therapy and the progression of the disease through radiological evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- HamadMC, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided